CLINICAL TRIAL: NCT06902740
Title: PCSK9 Inhibitor With Statin Therapy for Asymptomatic Intracranial Atherosclerosis (PISTIAS-2): A Multicenter, Open-label, Blinded-endpoint, Randomized Controlled Trial
Brief Title: PCSK9 Inhibitor With Statin Therapy for Asymptomatic Intracranial Atherosclerosis
Acronym: PISTIAS-2
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Chinese PLA General Hospital (Other); Hebei General Hospital (Other); Taihe Hospital (Other); Weifang People's Hospital (Other); Nanjing First Hospital, Nanjing Medical University (Other); Baotou Central Hospital (Other); Jining First People's Hospital (Other); Liaocheng People's Hospital (Other); Tangshan Worker's Hospital (Other); Chongqing General Hospital (Other); First Affiliated Hospital of Harbin Medical University (Other); Cangzhou Hospital of Integrated Traditional Chinese and Western Medicine (Other); The First Affiliated Hospital of Zhengzhou University (Other); The Affiliated Hospital of Qingdao University (Other); Zhongnan Hospital (Other); Huashan Hospital (Other)
Responsible Party: Principal Investigator, Wei-Hai Xu, MD & PhD, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: I-24PJ2601; 2024ZD0521605 (Other Grant/Funding Number: the Noncommunicable Chronic Diseases-National Science and Technology Major Project); 82025013 (Other Grant/Funding Number: the National Science Fund for Distinguished Young Scholars)
Record Dates: First submitted 2025-03-16; First posted 2025-03-30 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Intracranial Atherosclerosis; Intracranial Artery Stenosis; Atherosclerotic Plaque
Keywords: Intracranial Atherosclerosis; intracranial artery stenosis; atherosclerotic plaque; high-resolution magnetic resonance imaging; PCSK9 inhibitor; statin; Recaticimab
MeSH Terms: conditions — Intracranial Arteriosclerosis; Plaque, Atherosclerotic | interventions — Hydroxymethylglutaryl-CoA Reductase Inhibitors

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Recaticimab plus Statin Group (Experimental): Recaticimab (450mg every 12 weeks subcutaneously) combined with rosuvastatin 10mg qn or atorvastatin 20mg qn
  Interventions: Drug: Recaticimab and Statin
- Statin Group (Active Comparator): Rosuvastatin 10mg qn or atorvastatin 20mg qn
  Interventions: Drug: Statin

INTERVENTIONS:
Drug: Recaticimab and Statin — Recaticimab (450mg every 12 weeks subcutaneously) combined with rosuvastatin 10mg qn or atorvastatin 20mg qn
  Arms: Recaticimab plus Statin Group
Drug: Statin — Rosuvastatin 10mg qn or atorvastatin 20mg qn
  Arms: Statin Group

SUMMARY:
This is a prospective, multicenter, open-label, blinded-endpoint, randomized controlled trial designed to evaluate the efficacy and safety of PCSK9 inhibitor combined with statin therapy compared to statin monotherapy in reversing asymptomatic intracranial atherosclerosis, assessed using high-resolution magnetic resonance imaging of the intracranial vessel walls.

DETAILED DESCRIPTION:
Intracranial atherosclerotic stenosis (ICAS) is a leading cause of ischemic stroke worldwide, accounting for approximately 10-20% of all ischemic strokes in Europe and the United States, and up to 50% in Asian populations. While evidence-based management strategies for symptomatic ICAS have been progressively established over the past decades, asymptomatic ICAS - representing an earlier-stage, broader, high-risk population - has long been under-recognized and under-studied. Asymptomatic ICAS (stenosis > 50%) has a reported prevalence of approximately 6%-13%, and is associated with a substantially increased risk of future cerebrovascular events. Moreover, accumulating evidence has demonstrated that asymptomatic ICAS is independently associated with cognitive decline and incident dementia, likely due to chronic downstream hypo-perfusion and cumulative ischemic injury. Therefore, the development of systematic, evidence-based, and precision prevention strategies for asymptomatic ICAS is essential for reducing the overall disease burden attributable to ICAS-related cerebrovascular and neurodegenerative disorders.

It is well established that dysregulation of lipid metabolism is a fundamental pathophysiological mechanism driving the initiation and progression of ICAS, and low-density lipoprotein cholesterol (LDL-C) has been consistently identified as the primary therapeutic target for atherosclerotic cardiovascular disease and for the prevention of ischemic stroke. Existing evidence has demonstrated that reductions in lipid levels and the regression of atherosclerotic plaques are closely associated with a decreased risk of cardiovascular events. Statin therapy remains the cornerstone of lipid-lowering treatment, capable of stabilizing atherosclerotic plaques and improving clinical outcomes. However, limitations of statins such as the plateau effect of LDL-C reduction, intolerance, and poor adherence in certain patients necessitate alternative or adjunctive lipid-lowering strategies. Proprotein convertase subtilisin/kexin type 9 (PCSK9) inhibitors, human monoclonal antibodies targeting PCSK9, have shown excellent efficacy in achieving intensive LDL-C reduction and have been extensively validated for safety in large clinical trials. Recently published studies have highlighted the potential of PCSK9 inhibitors in plaque regression and stabilization beyond coronary and carotid arteries. The SLICE-CEA CardioLink-8 trial demonstrated that adding evolocumab to moderate- or high-intensity statin therapy for 6 months significantly reduced the lipid-rich necrotic core in asymptomatic high-risk carotid plaques. Similarly, the ARCHITECT study revealed that alirocumab in combination with high-intensity statin therapy led to significant regression of coronary plaque burden and enhanced plaque stability in asymptomatic patients over a 78-week period. Several observational studies have indicated that intensive lipid-lowering therapy may reverse asymptomatic ICAS. However, to date, no clinical trials have specifically evaluated the efficacy and safety of PCSK9 inhibitors in addition to statin therapy in patients with asymptomatic ICAS. This represents a critical evidence gap, as these patients constitute a broader, earlier, and high-risk population for cerebrovascular events.

The PISTIAS-2 is an investigator-initiated, multicentre, prospective, open-label, blinded end-point, randomized controlled trial designed to evaluate the efficacy and safety of PCSK9 inhibitor combined with statin therapy compared to statin monotherapy in patients with asymptomatic ICAS. Patients aged 18 to 60 years with asymptomatic ICAS, defined as 50% to 99% stenosis in at least one major intracranial artery without a prior history of ischemic stroke or transient ischemic attack, will be enrolled for 24-week treatment. Eligible participants will be centrally randomized into two groups: (1) Experimental group [PCSK9 inhibitor combined with statin therapy]: Recaticimab 450 mg every 12 weeks combined with rosuvastatin 10 mg q.n. or atorvastatin 20 mg q.n. (2) Control group [Statin alone]: Rosuvastatin 10 mg q.n. or atorvastatin 20 mg q.n. Considering inter-individual variability in lipid-lowering response, ezetimibe 10 mg once daily is permitted at the discretion of the study physician based on the predefined criteria: (1) patients already receiving statin therapy prior to enrollment whose LDL-C remains above 2.6 mmol/L, and (2) statin-naïve patients whose LDL-C exceeds 2.6 mmol/L at the 12-week lipid profile reassessment. In this trial, we employed a novel PCSK9 inhibitor, Recaticimab, a humanized IgG1 monoclonal antibody engineered with a strategic YTE mutation in its Fc region, which enhances its affinity for the neonatal Fc receptor (FcRn). This modification reduces FcRn-mediated antibody catabolism, thereby extending the half-life of Recaticimab and enabling a prolonged dosing interval of up to 12 weeks.

The primary outcome is the change in intracranial plaque burden from baseline to week 24, measured by high-resolution magnetic resonance imaging (HR-MRI).The key secondary outcomes include: change in stenosis degree from baseline to week 24, time from randomization to the first-ever ischemic stroke or transient ischemic attack, and change in plasma marker glial fibrillary acidic protein(GFAP) and neurofilament light (NfL). Other secondary outcomes include: time from randomization to the occurrence of major adverse cardiovascular events, new-onset silent cerebral infarction, percentage of patients who achieved LDL-C goal at week 24, percentage change in LDL-C relative to baseline, and change in plasma marker Aβ40, Aβ42, Aβ42/Aβ40. In addition, several pre-specified exploratory outcomes have been defined for this study. Details are provided in the "Outcome Measures" section.

After the 24-week treatment period, an extended prospective follow-up (clinical or telephone follow-up) will continue for more than one year to document long-term effects.The sample size is calculated based on the primary outcome and a total of 300 participants are anticipated. An interim analysis will be conducted when 50% of the participants (i.e., 150 subjects) have completed the 24-week follow-up with HR-MRI. An independent Data Safety Monitoring Board will oversee the overall conduct of the trial.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 and ≤60, male or female;
2. Asymptomatic intracranial artery stenosis (50%-99%) in the internal carotid artery (C6-7 segments), middle cerebral artery (M1 segment), vertebral artery (V4 segment), or basilar artery, confirmed by angiography (MRA, CTA, or DSA);
3. Atherosclerosis identified as the cause of intracranial artery stenosis by high-resolution magnetic resonance imaging;
4. No previous ischemic cerebrovascular events (including ischemic stroke or transient ischemic attack).
5. Baseline low-density lipoprotein cholesterol ≥ 2.6 mmol/L;
6. Informed consent signed.

Exclusion Criteria:

1. Non-atherosclerotic intracranial artery stenosis, including arterial dissection; moya moya disease; systemic vasculitis and primary central nervous system vasculitis; varicella-zoster vasculopathy or other viral vasculopathy; neurosyphilis and other intracranial infections, radiation vasculopathy; fibromuscular dysplasia, sickle cell disease, neurofibromatosis; reversible cerebral vasoconstriction syndrome; postpartum vasculopathy; suspected vasospasm, suspected reperfusion after vessel occlusion.
2. Upstream tandem extracranial vessel stenosis (≥50%) adjacent to the target intracranial stenotic vessel.
3. Previous treatment of target intracranial lesion with endovascular intervention or plan to perform endovascular intervention within 6 months, including intracranial stenting, endovascular angioplasty, and thrombectomy.
4. Any intracranial hemorrhage (parenchymal, subarachnoid, subdural, extradural, intraventricular) within 90 days prior to enrollment.
5. Presence of intracranial tumors.
6. Presence of cerebral aneurysms or arteriovenous malformations with indications for interventional therapy.
7. Major surgery (including open femoral, aortic, or carotid surgery) within previous 30 days or planned in the next 6 months after enrollment.
8. Presence of any of the following unequivocal cardiac sources of embolism: mitral stenosis, mechanical valve, endocarditis, intracardiac clot or vegetation, myocardial infarction within 3 months, dilated cardiomyopathy, chronic or paroxysmal atrial fibrillation.
9. New York Heart Association (NYHA) class III or IV, or known left ventricular ejection fraction < 30%.
10. Severe liver dysfunction or severe kidney dysfunction: AST and/or ALT > 3 times the ULN; creatinine clearance < 0.6 mL/s and/or serum creatinine > 265 μmol/L (>3.0 mg/dL); CK >5 times the ULN at screening.
11. Active bleeding diathesis or coagulopathy (e.g., active peptic ulcer disease, major systemic hemorrhage within 30 days, active bleeding diathesis, platelets count < 125,000 / uL, hematocrit < 30%, Hgb < 10 g/dl, international normalized ratio >1.5, bleeding time > 1 minute beyond normal value upper limit).
12. Presence of systemic autoimmune diseases: systemic sclerosis, systemic lupus erythematosus, Sjögren's syndrome, Behçet's disease, mixed connective tissue disease, IgG4-related disease.
13. Dementia or psychiatric problem that hinder their ability to consistently adhere to an outpatient program. Co-morbid conditions that may limit the life expectancy to less than 3 years.
14. Relative/absolute contraindications to magnetic resonance imaging (MRI) (such as presence of internal metallic objects, claustrophobia, contrast agent allergy, severe renal impairment, epilepsy, hypotension, asthma, and other hypersensitivity respiratory diseases).
15. Uncontrolled hypertension during the screening period, defined as seated systolic blood pressure (SBP) > 180 mmHg or diastolic blood pressure (DBP) > 110 mmHg.
16. Prior use of PCSK9 inhibitor before this recruitment.
17. Known intolerance or allergy to statin.
18. Pregnancy, lactation, or planning pregnancy.
19. Currently participating in another study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in plaque burden from baseline to week 24 | From baselie to the end of treatment at 24 weeks
  Intracranial plaque burden was assessed at maximum stenosis site by high-resolution magnetic resonance imaging, performed at baseline and the end of the treatment period (24 [±1] week) on the same machine. The plaque burden is calculated according to the following formula: plaque burden = [(vessel wall cross-sectional area - lumen cross-sectional area ) / vessel wall cross-sectional area] ×100%. The outcome will be centrally assessed by an independent core imaging laboratory blinded to treatment allocation according to a predefined imaging analysis protocol.

SECONDARY OUTCOMES:
Change in stenosis degree from baseline to week 24 | From baseline to the end of treatment at 24 weeks
  The degree of stenosis is calculated according to the Warfarin-Aspirin Symptomatic Intracranial Disease (WASID) criteria using the formula: [1-(Dstenosis/Dnormal)]×100%. Dstenosis represents the vessel diameter at the most stenotic site of the intracranial artery, and Dnormal represents the normal vessel diameter at a reference site.
Time from randomization to the first-ever ischemic stroke or transient ischemic attack | From baseline to the end of treatment at 24 weeks
  Ischemic Stroke: Defined as an acute cerebral infarction with clinical signs or imaging evidence of a new acute focal neurological injury persisting for more than 24 hours, excluding other non-ischemic causes.
  Transient Ischemic Attack (TIA): Defined as a sudden onset of focal neurological deficit due to cerebral or retinal ischemia, which completely resolves within 24 hours. Imaging (CT or MRI) must show no evidence of a new cerebral infarction. Other non-ischemic causes, such as brain infection, trauma, tumor, epilepsy, severe metabolic disorders, or progressive neurological diseases, must be excluded.
Change in plasma marker glial fibrillary acidic protein(GFAP) | From baseline to the end of treatment at 24 weeks
  Change in plasma marker glial fibrillary acidic protein(GFAP) quantified using the Single Molecule Array platform from baseline to the end of treatment at 24 weeks
Change in plasma marker neurofilament light(NfL) | From baseline to the end of treatment at 24 weeks
  Change in plasma marker Neurofilament light(NfL) quantified using the Single Molecule Array platform from baseline to the end of treatment at 24 weeks
Time from randomization to the occurrence of major adverse cardiovascular events | From baseline to the end of treatment at 24 weeks
  Composite major adverse cardiovascular endpoints includes ischemic stroke, myocardial infarction, and cardiovascular mortality as a cluster
Silent cerebral infarction | at 24 weeks of treatment
  New-onset silent cerebral infarction is defined as an imaging-detected infarct without acute clinical symptoms
Percentage of patients who achieved LDL-C goal at week 24 | at 24 weeks of treatment
  Percentage of patients achieving the LDL-C target at week 24 of treatment, defined as LDL-C < 1.8 mmol/L or LDL-C < 2.6 mmol/L based on ASCVD risk assessment.
Percentage change in LDL-C relative to baseline | From baseline to the end of treatment at 24 weeks
  Percentage change in LDL-C level at 24 weeks of treatment relative to baseline
Change in Plasma marker Aβ42/Aβ40 | From baseline to the end of treatment at 24 weeks
  Change in plasma markers Aβ42/Aβ40 from baseline to the end of treatment at 24 weeks

OTHER OUTCOMES:
Time from randomization to the time of the first occurrence of transient ischemic attack | From baseline to the end of treatment at 24 weeks
  Transient Ischemic Attack (TIA): Defined as a sudden onset of focal neurological deficit due to cerebral or retinal ischemia, which completely resolves within 24 hours. Imaging (CT or MRI) must show no evidence of a new cerebral infarction. Other non-ischemic causes, such as brain infection, trauma, tumor, epilepsy, severe metabolic disorders, or progressive neurological diseases, must be excluded.
Time from randomization to the time of the first occurrence of ischemic stroke | From baseline to the end of treatment at 24 weeks
  Ischemic Stroke: Defined as an acute cerebral infarction with clinical signs or imaging evidence of a new acute focal neurological injury persisting for more than 24 hours, excluding other non-ischemic causes.
Time from randomization to the time of the occurrence of any stroke | From baseline to the end of treatment at 24 weeks
  Any stroke includes ischemic and hemorrhagic stroke
Time from randomization to the time of the occurrence of myocardial infarction | From baseline to the end of treatment at 24 weeks
  Time from randomization to the time of the occurrence of myocardial infarction
Time from randomization to the time of the occurrence of vascular death | From baseline to the end of treatment at 24 weeks
  Time from randomization to the time of the occurrence of vascular death
Time from randomization to the time of the occurrence of any death | From baseline to the end of treatment at 24 weeks
  All-cause mortality will be calculated between two arms
Changes in cognitive scale scores | From baseline to the end of treatment at 24 weeks
  Cognitive function will be evaluated via MMSE and MOCA at baseline and week 24
Changes in traditional lipid parameters | From baseline to the end of treatment at 24 weeks
  Changes in traditional lipid profiles, especially total cholesterol (TC), triglycerides (TG) and HDL-C.
Change in Lipoprotein (a) level | From baseline to the end of treatment at 24 weeks
  Non-traditional lipid parameters such as Lipoprotein (a) level will be detected at baseline and week 24
Visit-to-visit lipid variability of LDL-C | From baseline to the end of treatment at 24 weeks
  Lipid variability during the treatment period, which can be evaluated by the following indicators: coefficient of variation (CV), standard deviation (SD), variability independent of the mean (VIM), average real variability (ARV).
Change in high-sensitivity C-reactive protein | From baseline to the end of treatment at 24 weeks
  Inflammatory markers such as high-sensitivity C-reactive protein (hs-CRP) will be detected at baseline and week 24
Change in plasma marker pTau217 | From baseline to the end of treatment at 24 weeks
  Markers of neurological disorders such asplasma marker pTau217 will be detected at baseline and week 24
Changes in DNA methylation status of peripheral blood cells | From baseline to the end of treatment at 24 weeks
  DNA methylation, particularly RNF213, an important epigenetic factor, may play a role in the progression of ICAS.
Changes in Senescence-Associated Secretory Phenotype | From baseline to the end of treatment at 24 weeks
  Previous studies have shown that lipid-lowering has an obvious scavenging effect on senescent cells. Senescence associated β-galactosidase, SA-β-gal, is thought to be a sign of aging
Change in length of plaque | From baseline to the end of treatment at 24 weeks
  length of plaque was evaluated by high-resolution MRI at baseline and week 24
Change in plaque maximum thickness | From baseline to the end of treatment at 24 weeks
  the maximum thickness of plaque was evaluated by high-resolution MRI at baseline and week 24
Change in the outer-wall boundary area at the maximal stenotic site | From baseline to the end of treatment at 24 weeks
  the outer-wall boundary area at the maximal stenotic site was evaluated by high-resolution MRI at baseline and week 24
Change in remodeling index of the plaque | From baseline to the end of treatment at 24 weeks
  Remodeling index of the plaque is calculated by the ratio of the diameter of the lumen at the most severe lesion to the diameter of the proximal reference lumen, positive remodeling defined as remodeling index > 1.1
Change in plaque enhancement | From baseline to the end of treatment at 24 weeks
  plaque enhancement will be detected via contrast enhanced high- resolution MRI
Change in brain volume | From baseline to the end of treatment at 24 weeks
  Total brain volume will be evaluated by MRI 3D-T1WI at baseline and week 24
Change in cortical thickness | From baseline to the end of treatment at 24 weeks
  The thickness and surface area of cerebral cortex in all and different brain regions were quantitatively determined based on MRI
Change in cerebral small vessel disease burden | From baseline to the end of treatment at 24 weeks
  cerebral small vessel disease burden were quantitatively determined based on MRI at baseline and week 24
Change in white matter hyperintensity | From baseline to the end of treatment at 24 weeks
  White matter hyperintensity (WMH) in all and different brain regions were quantitatively determined based on MRI
Change in collateral circulation status | From baseline to the end of treatment at 24 weeks
  Collateral circulation status will be assessed using standardized imaging-based grading scales to evaluate the extent and quality of collateral blood flow.
Adverse events | From baseline to the end of treatment at 24 weeks
  An Adverse Event (AE) is any untoward medical occurrence in clinical trial subject administered a pharmaceutical product and which does not necessarily have a causal relationship with the treatment.
Serious Adverse Events | From baseline to the end of treatment at 24 weeks
  A Serious Adverse Event (SAE) is any untoward medical occurrence that, at any dose: (1) results in death; (2) is life-threatening; (3) requires inpatient hospitalization or prolongation of existing hospitalization; (4)results in persistent or significant disability/incapacity; (5) is a congenital anomaly/birth defect; (6) is otherwise considered medically significant by the investigator.

CONTACTS AND LOCATIONS:
Locations (19):
- China (19):
  - Peking Union Medical College Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality
  - Chinese PLA General Hospital, Beijing, Beijing Municipality
  - The Third Affiliated Hospital of Sun Yat-sen University, Yuedong Hospital, Meizhou, Guangdong
  - Cangzhou Hospital of Integrated Traditional Chinese and Western Medicine, Cangzhou, Hebei
  - Peking University Third Hospital Qinhuangdao Hospital, Qinhuangdao, Hebei
  - Hebei Provincial People's Hospital, Shijiazhuang, Hebei
  - Tangshan Worker's Hospital, Tangshan, Hebei
  - First Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - The first affiliated hospital of zhengzhou university, Zhengzhou, Henan
  - Taihe Hospital, Shiyan, Hubei
  - Zhongnan Hospital of Wuhan University, Wuhan, Hubei
  - Baotou Central Hospital, Baotou, Inner Mongolia
  - Nanjing First Hospital, Nanjing, Jiangsu
  - Jining First People's Hospital, Jining, Shandong
  - Liaocheng People's Hospital, Liaocheng, Shandong
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Weifang People's Hospital, Weifang, Shandong
  - Chongqing General Hospital, Chongqing
  - Huashan Hospital, Fudan University, Shanghai

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Perez de Isla L, Diaz-Diaz JL, Romero MJ, Muniz-Grijalvo O, Mediavilla JD, Argueso R, Sanchez Munoz-Torrero JF, Rubio P, Alvarez-Banos P, Ponte P, Manas D, Suarez Gutierrez L, Cepeda JM, Casanas M, Fuentes F, Guijarro C, Angel Barba M, Saltijeral Cerezo A, Padro T, Mata P; SAFEHEART Study Group. Alirocumab and Coronary Atherosclerosis in Asymptomatic Patients with Familial Hypercholesterolemia: The ARCHITECT Study. Circulation. 2023 May 9;147(19):1436-1443. doi: 10.1161/CIRCULATIONAHA.122.062557. Epub 2023 Apr 3. PMID 37009731
- [Background] Sabatine MS, Giugliano RP, Keech AC, Honarpour N, Wiviott SD, Murphy SA, Kuder JF, Wang H, Liu T, Wasserman SM, Sever PS, Pedersen TR; FOURIER Steering Committee and Investigators. Evolocumab and Clinical Outcomes in Patients with Cardiovascular Disease. N Engl J Med. 2017 May 4;376(18):1713-1722. doi: 10.1056/NEJMoa1615664. Epub 2017 Mar 17. PMID 28304224
- [Background] Nicholls SJ, Puri R, Anderson T, Ballantyne CM, Cho L, Kastelein JJ, Koenig W, Somaratne R, Kassahun H, Yang J, Wasserman SM, Scott R, Ungi I, Podolec J, Ophuis AO, Cornel JH, Borgman M, Brennan DM, Nissen SE. Effect of Evolocumab on Progression of Coronary Disease in Statin-Treated Patients: The GLAGOV Randomized Clinical Trial. JAMA. 2016 Dec 13;316(22):2373-2384. doi: 10.1001/jama.2016.16951. PMID 27846344
- [Background] Kim BS, Lim JS, Jeong JU, Mun JH, Kim SH. Regression of asymptomatic intracranial arterial stenosis by aggressive medical management with a lipid-lowering agent. J Cerebrovasc Endovasc Neurosurg. 2019 Sep;21(3):144-151. doi: 10.7461/jcen.2019.21.3.144. Epub 2019 Sep 30. PMID 31886149
- [Background] Miao H, Yang Y, Wang H, Huo L, Wang M, Zhou Y, Hua Y, Ren M, Ren C, Ji X, Yang Q, Guo X. Intensive Lipid-Lowering Therapy Ameliorates Asymptomatic Intracranial Atherosclerosis. Aging Dis. 2019 Apr 1;10(2):258-266. doi: 10.14336/AD.2018.0526. eCollection 2019 Apr. PMID 31011477
- [Background] Zhu J, Wang Y, Li J, Deng J, Zhou H. Intracranial artery stenosis and progression from mild cognitive impairment to Alzheimer disease. Neurology. 2014 Mar 11;82(10):842-9. doi: 10.1212/WNL.0000000000000185. Epub 2014 Jan 31. PMID 24489130
- [Background] Zhao D, Guallar E, Qiao Y, Knopman DS, Palatino M, Gottesman RF, Mosley TH Jr, Wasserman BA. Intracranial Atherosclerotic Disease and Incident Dementia: The ARIC Study (Atherosclerosis Risk in Communities). Circulation. 2024 Sep 10;150(11):838-847. doi: 10.1161/CIRCULATIONAHA.123.067003. Epub 2024 Aug 1. PMID 39087353
- [Background] Gao P, Wang T, Wang D, Liebeskind DS, Shi H, Li T, Zhao Z, Cai Y, Wu W, He W, Yu J, Zheng B, Wang H, Wu Y, Dmytriw AA, Krings T, Derdeyn CP, Jiao L; CASSISS Trial Investigators. Effect of Stenting Plus Medical Therapy vs Medical Therapy Alone on Risk of Stroke and Death in Patients With Symptomatic Intracranial Stenosis: The CASSISS Randomized Clinical Trial. JAMA. 2022 Aug 9;328(6):534-542. doi: 10.1001/jama.2022.12000. PMID 35943472
- [Background] Chimowitz MI, Lynn MJ, Derdeyn CP, Turan TN, Fiorella D, Lane BF, Janis LS, Lutsep HL, Barnwell SL, Waters MF, Hoh BL, Hourihane JM, Levy EI, Alexandrov AV, Harrigan MR, Chiu D, Klucznik RP, Clark JM, McDougall CG, Johnson MD, Pride GL Jr, Torbey MT, Zaidat OO, Rumboldt Z, Cloft HJ; SAMMPRIS Trial Investigators. Stenting versus aggressive medical therapy for intracranial arterial stenosis. N Engl J Med. 2011 Sep 15;365(11):993-1003. doi: 10.1056/NEJMoa1105335. Epub 2011 Sep 7. PMID 21899409
- [Background] Li S, Tang M, Zhang D, Han F, Zhou L, Yao M, Li M, Cui L, Zhang S, Peng B, Jin Z, Zhu Y, Ni J. The prevalence and prognosis of asymptomatic intracranial atherosclerosis in a community-based population: Results based on high-resolution magnetic resonance imaging. Eur J Neurol. 2023 Dec;30(12):3761-3771. doi: 10.1111/ene.16057. Epub 2023 Sep 22. PMID 37738517
- [Background] Gutierrez J, Khasiyev F, Liu M, DeRosa JT, Tom SE, Rundek T, Cheung K, Wright CB, Sacco RL, Elkind MSV. Determinants and Outcomes of Asymptomatic Intracranial Atherosclerotic Stenosis. J Am Coll Cardiol. 2021 Aug 10;78(6):562-571. doi: 10.1016/j.jacc.2021.05.041. PMID 34353533
- [Background] Wong KS, Ng PW, Tang A, Liu R, Yeung V, Tomlinson B. Prevalence of asymptomatic intracranial atherosclerosis in high-risk patients. Neurology. 2007 Jun 5;68(23):2035-8. doi: 10.1212/01.wnl.0000264427.09191.89. PMID 17548555
- [Background] Wong KS, Huang YN, Yang HB, Gao S, Li H, Liu JY, Liu Y, Tang A. A door-to-door survey of intracranial atherosclerosis in Liangbei County, China. Neurology. 2007 Jun 5;68(23):2031-4. doi: 10.1212/01.wnl.0000264426.63544.ee. PMID 17548554